CLINICAL TRIAL: NCT00692666
Title: Letigen® and Cardiovascular Morbidity. A Register-Based Epidemiological Study
Brief Title: Letigen® and Cardiovascular Morbidity
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Nycomed Group, Langebjerg 1, 4000 Roskilde, Denmark (Unknown)
Responsible Party: Jesper Hallas, professor, University of Southern Denmark
Other Study IDs: Letigen
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Stroke; Myocardial Infarctions; Sudden Death
MeSH Terms: conditions — Stroke; Myocardial Infarction; Death, Sudden

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Letigen® was a combination drug containing ephedrine, an adrenergic agonist with lipolytic and appetite-inhibiting properties. The drug was used as adjuvant treatment of obesity from 1990 and up to 2002 when it was withdrawn from the market by the manufacturer. The basis for this was a number of spontaneous reports about patients that died during treatment with Letigen®.

The causal relation has never been addressed. There are only sparse data from randomised studies and the above-mentioned reports are not conclusive.

We propose a controlled study based on data from Statistics Denmark that hold a complete copy of the Prescription Register of the Danish Medicines Agency and the Danish Hospital Discharge Register. The aim of the study would be to determine whether there is an excess frequency of deaths and serious cardiovascular events that can not be explained by particular characteristics of users of the drug. A well-known problem in such observational studies is a fundamental incomparability between users and non-users of drugs. In the present setting, it should be expected that use of Letigen® is associated with high BMI, smoking, alcohol abuse, type-2 diabetes, mild hypertension, low physical activity and other indicators of unhealthy lifestyle. Thus, an uncritical comparison between users and non-users of Letigen® regarding serious cardiovascular events will probably show an excess frequency that can not necessarily be attributed to the drug. This problem can be addressed by a special epidemiological technique - the case-crossover design - which is particularly robust to such comparability problems. In brief, only cases should be included. Controls are the same persons at an earlier time, , where the case-defining disease has not yet developed. The exposure of cases will be compared with the exposure of the same persons' case history.

To account for the effect of chronic exposure, we also perform, as a secondary analysis, a conventional case-control study nested within the cohort of Letigen users, and employing a risk-set sampling technique.

ELIGIBILITY:
Inclusion Criteria:

* Use of letigen TM within the period Jan 1995 - Dec 2001
* The occurrence of a case-defining event

Exclusion Criteria:

* A cancer diagnosis other than non-melanoma skin cancer
* Age outside the range 18-70

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300000
Dates: Start 2006-05; Primary Completion 2006-05 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Hallas, Md PhD, Principal Investigator — University of Southern Denmark